CLINICAL TRIAL: NCT06947603
Title: Effect of Inula Viscosa Extract on Postoperative Bleeding and Healing After Lower Third Molar Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Wataniya University (Other)
Responsible Party: Principal Investigator, Tarek Khaled Abou Agwa, Senior lecturer, Al-Wataniya University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M/70- 14.10.2023
Record Dates: First submitted 2025-04-03; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Bleeding; Healing Surgical Wounds
Keywords: Inula Viscosa; Pain; Edema; Trismus; Lower Third Molars
MeSH Terms: conditions — Hemorrhage; Pain; Edema; Trismus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- inula viscosa extract was used for one side of patients after surgical lower third molar removal (Active Comparator): The study sample was divided into two equal groups based on the type of pharmaceutical substance applied within the alveolar socket after the extraction of impacted molars. In the first group (Inula group), an extract of INULA was used
  Interventions: Procedure: inula viscosa extract; Procedure: no inula viscosa extract
- nothing was used for other side of patients after surgical lower third molar removal (Active Comparator): The study sample was divided into two equal groups based on the type of pharmaceutical substance applied within the alveolar socket after the extraction of impacted molars. In the second group (control group), nothing was used
  Interventions: Procedure: inula viscosa extract; Procedure: no inula viscosa extract

INTERVENTIONS:
Procedure: inula viscosa extract — the topical gel of inula viscosa was applied to one side after the extraction of the impacted molar in each patient, while the other side was left without the application of any pharmaceutical substance after extraction
Procedure: no inula viscosa extract — the other side of patient was left without the application of inula viscosa extract after lower third molar extraction.

SUMMARY:
In oral surgery, the operation of the impacted third molar is one of the most common surgical procedures performed by oral and maxillofacial surgeons .Several attempts have been made to reduce the postoperative outcome of the removal of the third molar post-surgery.The bioactive components in Inula extracts consist of sesquiterpene lactones, and the major components are alantolactone and isoalantolactone .]. Inula has Antioxidant, antihyperglycemic, antimicrobial, antibacterial, antifungal, anticancer and anti-inflammatory effects. the purpose of this study was to assess the effects of inula viscosa on the postoperative period of the third molar surgery by evaluating bleeding, and healing.

DETAILED DESCRIPTION:
material and method: A total of 30 patients aged 18 to 35 years were enrolled in the study. The inclusion criteria for the study group were as follows: bilateral lower impacted third molars (those that can only be surgically extracted through bone osteotomy with or without the need for tooth sectioning) , non-smokers, good general health with no systemic diseases, not pregnant or lactating, no medication taken that could influence wound healing after surgery, and no oral inflammation, such as periodontal disease. The study sample was divided into two equal groups based on the type of pharmaceutical substance applied within the alveolar socket after the extraction of impacted molars. In the first group (Inula group), an extract of INULA was used, while in the second group (controlled group), nothing was used. In both groups, the pharmaceutical substance was applied to one side after the extraction of the impacted molar in each patient, while the other side was left without the application of any pharmaceutical substance after extraction. It is noteworthy that the second extraction on the patient was only performed after complete healing of the controlled side. Before the surgical procedure, each patient received information about the surgery, postoperative recommendations, and possible complications. They signed a consent form indicating their agreement to participate in the study. The study protocol and consent form were approved by Al-Wataniya Private University, Syria. after syrgery All patients received postoperative instructions.

Measurement of bleeding:

A subjective method was used to compare post-operative bleeding between the two techniques in this clinical trial. The patient was asked to count the number of gauze pads for the patient to bite on gauzes used to stop bleeding, for each surgical site, on each day post-operatively, also, the patient reported the time needed to achieve a bleeding-free surgical site measurement of post-operative healing:

The assessment of socket healing was carried out at one week after surgery using a five-grade index to measure the degree of socket epithelization, which was designed by (Alkadi 2018) as follows :

Healing grade

* Very poor (1) : Clinical criteria Tissue color: ˃ 50% of gingivae red , Response to palpation: bleeding, Granulation tissue: present, Incision margin: not epithelialized, with loss of epithelium , beyond margins .Suppuration: present
* Poor (2) : Tissue color:˃ 50% of gingivae red, Response to palpation: bleeding, Granulation tissue: present Incision margin: not epithelialized, with connective tissue exposed, Suppuration: none
* Good (3) : Tissue color: ˂ 50% of gingivae red, Response to palpation: no bleeding, Granulation tissue: none, Incision margin: no connective tissue exposed, Suppuration: none
* Very good (4) :Tissue color: ˂ 25% of gingivae red, Response to palpation: no bleeding, Granulation tissue: none, Incision margin: no connective tissue exposed, Suppuration: none
* Excellent (5) :Tissue color: all gingivae pink, Response to palpation: no bleeding, Granulation tissue: none, Incision margin: no connective tissue exposed, Suppuration: none Statistical analysis Recorded data were analyzed using the IBM SPSS 20.0 software (Statistical Package for the Social Science, SPSS Inc., Chicago, IL, USA).

ELIGIBILITY:
Inclusion Criteria:

* patients have bilateral lower impacted third molars (those that can only be surgically extracted through bone osteotomy with or without the need for tooth sectioning)
* good general health with no systemic diseases, ,

Exclusion Criteria:

* non-smokers,
* no medication taken that could influence wound healing after surgery,
* and no oral inflammation, such as periodontal disease,
* for woman not pregnant or lactating.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female participate has to be not pregnant or lactating
Enrollment: 30 (Actual)
Dates: Start 2023-11-20 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-29 (Actual)

PRIMARY OUTCOMES:
questionnaire | postprocedural, up to 12 hours
  Measurement of bleeding:
  A subjective method was used to compare post-operative bleeding between the two techniques in this clinical trial. The patient was asked to count the number of gauze pads for the patient to bite on gauzes used to stop bleeding, for each surgical site, on each day post-operatively, also, the patient reported the time needed to achieve a bleeding-free surgical site
healing after surgery as assessed by Alkadi 2018 | time 1: one week after surgery
  The assessment of socket healing was carried out at one week after surgery using a five-grade index to measure the degree of socket epithelization, which was designed by (Alkadi 2018) as follows :
  * Very poor (1) : Clinical criteria Tissue color: ˃ 50% of gingivae red , Response to palpation: bleeding, Granulation tissue: present, Incision margin: not epithelialized, with loss of epithelium , beyond margins .Suppuration: present
  * Poor (2) : Tissue color:˃ 50% of gingivae red, Response to palpation: bleeding, Granulation tissue: present Incision margin: not epithelialized, with connective tissue exposed, Suppuration: none
  * Good (3) : Tissue color: ˂ 50% of gingivae red, Response to palpation: no bleeding, Granulation tissue: none, Incision margin: no connective tissue exposed, Suppuration: none
  * Very good (4) :Tissue color: ˂ 25% of gingivae red, Response to palpation: no bleeding, Granulation

CONTACTS AND LOCATIONS:
Locations (1):
- Al Wataniya Private University, Hama, Hama Government, Syria

IPD SHARING:
Plan to Share IPD: No